CLINICAL TRIAL: NCT05109065
Title: Peripheral Immune System in Individuals With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Agnieszka Kalinowski, Clinical Asst Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 58926
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Schizophreniform Disorders
Keywords: psychosis; psychiatry; complement immune system
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators want to save private information and/or specimens for future research. The study collects 5 Tablespoons of blood. As part of the analysis on your specimens, the investigators may do genetic testing. Genetic research is research that studies genes, including gene characteristics and gene versions that are transmitted by parents to children. Your specimens will be stored using an assigned study code number and unlinked to your identifying information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with primary psychotic disorders: Participants who have received any of the following diagnoses: schizophrenia, schizoaffective disorder, or schizophreniform disorder.
  Participants will have urine toxicology screen, vitals recorded, and blood drawn in a single visit.
  Interventions: Diagnostic Test: SCID (Standardized Clinical Interview for DSM-V); Diagnostic Test: PSS (Perceived Stress Score); Diagnostic Test: Urine Toxicology Screen; Diagnostic Test: Vitals; Diagnostic Test: Blood Work; Diagnostic Test: COVID Screening; Diagnostic Test: Positive and Negative Syndrome Scale (PANSS)
- Healthy Controls: Healthy participants who do not have any exclusion criteria will undergo an assessment to confirm absence of psychiatric disorder.
  Participants will have urine toxicology screen, vitals recorded, and blood drawn in a single visit.
  Interventions: Diagnostic Test: SCID (Standardized Clinical Interview for DSM-V); Diagnostic Test: PSS (Perceived Stress Score); Diagnostic Test: Urine Toxicology Screen; Diagnostic Test: Vitals; Diagnostic Test: Blood Work; Diagnostic Test: PQ-B; Diagnostic Test: COVID Screening

INTERVENTIONS:
Diagnostic Test: SCID (Standardized Clinical Interview for DSM-V) — The Structured Clinical Interview for DSM-5 (SCID-5) is a semistructured interview guide for a clinician or trained mental health professional to diagnose major mental illnesses.
Diagnostic Test: PSS (Perceived Stress Score) — The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. Demographic information will also be collected.
Diagnostic Test: Urine Toxicology Screen — Participants will be asked to provide a urine sample. Evidence of active substance abuse (marijuana, opioids, other non-prescription drugs) by the urine toxicology screen will disqualify participants from the study.
Diagnostic Test: Vitals — Height and weight will be measured in order to calculate BMI.
Diagnostic Test: Blood Work — A venipuncture will be performed for the purpose of collecting blood tissue for study.
Diagnostic Test: PQ-B — The Prodromal Questionnaire - Brief Version (PQ-B) is a self-report measure designed to identify people who may be experiencing psychotic symptoms when they do not have a schizophrenia diagnosis.
  Groups: Healthy Controls
Diagnostic Test: COVID Screening — Questionnaire to assess risk of transmission of COVID-19.
Diagnostic Test: Positive and Negative Syndrome Scale (PANSS) — Instrument that is completed by clinical interviewer to measure symptom severity in individuals with psychotic disorders.
  Groups: Individuals with primary psychotic disorders

SUMMARY:
The investigators are seeking healthy volunteers and people with schizophrenia or schizoaffective disorder for a clinical study of the immune system in psychotic disorders. This is an observational study, to understand the ways in which the immune system may be contributing to the disease process.

DETAILED DESCRIPTION:
Genetic studies have linked the number of copies coding for C4 protein to risk for schizophrenia. Studies examining the amount of mRNA, the molecules that point to how much C4 protein is likely being made, found more C4 mRNA in the brains from individuals with schizophrenia. Studies in mice have suggested that expressing more C4 protein in the brain, specifically the A-type of C4, can result in abnormalities in behavior. However, researchers have also found that pathways that involve this protein in the blood to be abnormal in individuals even before they develop schizophrenia and hypothesize these abnormalities change the blood brain barrier. In this work, the researchers are hoping to understand the ways in which C4 protein is abnormal in the peripheral blood and how this may be contributing to the disease process in hopes of finding new ways of helping individuals with schizophrenia and possibly other mental health disorders. A major goal of this study is to collect blood tissue for ongoing translational study of pathophysiological mechanisms of schizophrenia.

Interested participants will be asked a series of questions about their medical and mental health history, be able to provide informed consent, undergo a urine toxicology screen and be willing to provide a blood sample.

ELIGIBILITY:
Inclusion Criteria for Subjects with schizophrenia and schizoaffective disorders:

* Schizophrenia or schizoaffective disorder diagnosis verified by interview
* Diagnosis or initiation of antipsychotic medication was within last 5 years

Inclusion Criteria for Healthy Controls:

* No known diagnosis of schizophrenia or schizoaffective disorder
* No history of depression, anxiety, bipolar disorder, PTSD, agoraphobia, panic disorder, or generalized anxiety disorder
* Negative assessment for psychotic symptoms on day of interview

Exclusion Criteria (for both groups):

* Participants have a history of bleeding disorders or are taking blood thinners.
* Participants have a history of epilepsy, known genetic disorders
* Immunocompromised state (eg., receiving immunosuppressive therapy, transplant).
* History of brain-related disease (eg., stroke)
* Any uncontrolled medical disorder such as cancer.
* History of substance abuse or positive urine toxicology screen (including test for marijuana) on the day of the blood draw

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients seen at local outpatient clinics for schizophrenia, local community residents, and volunteers on clinical study database.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Group comparison of C4 protein in immune cells | Day 1
  Measure the concentration of complement 4 protein in immune cells.

SECONDARY OUTCOMES:
Body Mass Index and its relationship to C4 protein concentration | Day 1
  The relationship between body mass index, calculated from the measured height and weight of participants, and the primary outcome (C4 protein concentration) will be determined.
C4 Gene Copy Number | Day 1
  Determine the C4 Gene Copy Number its relationship to C4 protein concentration in immune cells.
C4 Activation | Day 1
  Measure activity of C4 protein and its relationship to the primary outcome.
Relationship to symptom presentation | Day 1
  Explore the relationship between clinical severity scores (PANSS) and the primary outcome.
Relationship to stress | Day 1
  Explore the relationship between perceived stress (PSS) and the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Kalinowski, MD PhD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Background] Kalinowski A, Liliental J, Anker LA, Linkovski O, Culbertson C, Hall JN, Pattni R, Sabatti C, Noordsy D, Hallmayer JF, Mellins ED, Ballon JS, O'Hara R, Levinson DF, Urban AE. Increased activation product of complement 4 protein in plasma of individuals with schizophrenia. Transl Psychiatry. 2021 Sep 22;11(1):486. doi: 10.1038/s41398-021-01583-5. PMID 34552056
- See also: Laskaris, et.al. Schizophr Res . 2019 Feb;204:30-37. — https://pubmed.ncbi.nlm.nih.gov/30527272/
- See also: Yilmaz, et. al. Nat Neurosci . 2021 Feb;24(2):214-224. — https://www.nature.com/articles/s41593-020-00763-8
- See also: Sekar, at al. Nature . 2016 Feb 11;530(7589):177-83. — https://pubmed.ncbi.nlm.nih.gov/26814963/
- See also: Radhakrishnan, et al. Mol Psychiatry . 2021 Jun 16. — https://www.nature.com/articles/s41380-021-01184-0
- See also: Onwordi, et. al. Transl Psychiatry . 2021 Jul 17;11(1):393. — https://www.nature.com/articles/s41398-021-01515-3
- See also: Onwordi, et. al. Nat Commun . 2020 Jan 14;11(1):246. — https://www.nature.com/articles/s41467-019-14122-0

DOCUMENTS (1):
  • Informed Consent Form (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT05109065/ICF_001.pdf